CLINICAL TRIAL: NCT01211314
Title: Treatment of Essential Hypertension With Vasodip-Combo 20. Efficacy and Safety Evaluation With 24 h Ambulatory Blood Pressure Measurements
Brief Title: Antihypertensive Efficacy of Fixed Combination Drug
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Meir Medical Center (Other)
Collaborators: Dexcel Pharma Technologies Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDU1952
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2011-08

CONDITIONS: Hypertension
Keywords: hypertension; Fixed combination; lercanidipine; enalapril; Blood Pressure Monitoring, Ambulatory
MeSH Terms: conditions — Hypertension | interventions — lercanidipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lercanidipine-enalapril fixed combination (Experimental): uncontrolled hypertensive patients will receive fixed combination therapy
  Interventions: Drug: Lercanidipine/enalapril fixed combination

INTERVENTIONS:
Drug: Lercanidipine/enalapril fixed combination — Lercanidipine 10 mg + enalapril 20 mg, once a day, used as a fixed combination drug. Unique dose during the study
  Other Names: Vasodip Combo 20; hypertension; ambulatory blood pressure monitoring

SUMMARY:
Treatment and control of hypertension is still insufficient. About 50% of the patients remain uncontrolled. Lack of compliance with discontinuation of drug treatment is an important reason for not achieving blood pressure. Several studies have shown that use of fixed combinations improve compliance significantly, by reducing the number of pill's intake.

This study will assess the antihypertensive efficacy of Vasodip-Combo 20® [enalapril 20 mg + lercanidipine 10 mg] as a fixed combination drug in uncontrolled antihypertensive patients.

DETAILED DESCRIPTION:
This is a single centre observational uncontrolled prospective study, Hypertensive patients that are either treatment naïve or uncontrolled on current therapy [one or two drugs] and meet all inclusion and exclusion criteria, will be assigned to Vasodip-Combo 20 as unique drug treatment. The treatment will then be continued for additional 4 weeks. Office blood pressure will be performed by the physician at each visit. 24 h. ambulatory blood pressure measurements [ABPM] and blood samples for electrolytes, creatinine and urea will be taken at base line visit and at at week 4.

Efficacy will be defined in terms of therapeutic goals expressed as target blood pressures according to World Health Organization and European society of Hypertension [ for office blood pressure and ambulatory blood pressure measurements] criteria:

Office Blood Pressure: Diastolic blood pressure ≤ 90 mmHg and Systolic blood pressure ≤ 140 mmHg for non-diabetics or Diastolic Blood Pressure ≤ 80 mmHg and Systolic Blood Pressure ≤ 130 mmHg for diabetics, respectively.

24 h Ambulatory Blood Pressure Measurements: 224 Hour: Diastolic Blood Pressure≤ 80 mmHg and Systolic Blood Pressure ≤ 130 mmHg, Awake time: Diastolic Blood Pressure ≤ 85 mmHg,Systolic Blood Pressure ≤ 135 mmHg Asleep Time: Diastolic Blood Pressure ≤70 mmHg, Systolic Blood Pressure ≤ 70 mmHg.

Effectiveness and Safety will also be evaluated taking into consideration patient compliance

Safety assessments:

Safety will be assessed by means of (S)Adverse effects reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension at visit 1 defined as office blood pressure <140/90 mmHg and a 24 h ABPM >130/80 mmHg with a day time blood pressure (extracted from the 24h ABPM) >135/85 mmHg
2. Male and female
3. Age 18-80
4. Every patient that in the medical opinion of the treating physician is eligible for Vasodip Combo 20 treatment.
5. Willing to sign an informed consent

Exclusion Criteria:

1. Use of more than 2 anti hypertensive medication at visit 1 (fixed combination is considered as two drugs)
2. Mean 24 h ABPM values of more than 180/100 mmHg
3. Pregnant women
4. Women with potential age of pregnancy.
5. Suspected secondary hypertension (investigator decision)
6. Uncontrolled Diabetes Mellitus(investigator decision)
7. Any of the following in the last six months: Myocardial Infarction, Stroke, Coronary by-pass surgery, Percutaneous coronariography with balloon dilation and/or stent insertion
8. Congestive Heart Failure requiring pharmacological treatment
9. Renal Failure, defined as serum creatinine equal or great than 1.5 mg% [confirmed twice] or hyperkalemia defined as serum potassium equal or great that 5 meq/l [confirmed twice]
10. Malignancy that required Chemotherapy in the last 3 years.
11. Any medical or none medical condition that in the eyes of the investigator will not allow the patient to complete the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Blood Pressure control | Four weeks
  Percentage of patients with controlled blood pressure with office BP and 24 h ABPM measurements, from baseline to week 4.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Podjarny, MD, Principal Investigator — Clalit Health Services
Locations (1):
- Clalit Health Services, Herzliya, Hasharon, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hair PI, Scott LJ, Perry CM. Fixed-dose combination lercanidipine/enalapril. Drugs. 2007;67(1):95-106; discussion 107-8. doi: 10.2165/00003495-200767010-00007. PMID 17209666
- [Background] Menne J, Haller H. Fixed-dose lercanidipine/enalapril for hypertension. Drugs Today (Barc). 2008 Apr;44(4):261-70. doi: 10.1358/dot.2008.44.4.1164756. PMID 18536784
- [Background] Mancia G, Laurent S, Agabiti-Rosei E, Ambrosioni E, Burnier M, Caulfield MJ, Cifkova R, Clement D, Coca A, Dominiczak A, Erdine S, Fagard R, Farsang C, Grassi G, Haller H, Heagerty A, Kjeldsen SE, Kiowski W, Mallion JM, Manolis A, Narkiewicz K, Nilsson P, Olsen MH, Rahn KH, Redon J, Rodicio J, Ruilope L, Schmieder RE, Struijker-Boudier HA, Van Zwieten PA, Viigimaa M, Zanchetti A. Reappraisal of European guidelines on hypertension management: a European Society of Hypertension Task Force document. Blood Press. 2009;18(6):308-47. doi: 10.3109/08037050903450468. No abstract available. PMID 20001654